CLINICAL TRIAL: NCT00991341
Title: Red Cell Storage Duration Study
Acronym: RECESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 676; U01HL072268 (NIH); HL072268; HL072033; HL072291; HL072196; HL072289; HL072248; HL072191; HL072299; HL072305; HL072274; HL072028; HL072359; HL072072; HL072355; HL072283; HL072346; HL072331; HL072290
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2014-05

CONDITIONS: Cardiac Surgery; Erythrocyte Transfusion
Keywords: Cardiac surgery; Red blood cell; Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shorter-storage red blood cell units (Active Comparator): Red blood cell units stored <= 10 days
  Interventions: Biological: Red blood cell units stored <= 10 days
- Longer-storage red blood cell units (Active Comparator): Red blood cell units stored >= 21 days
  Interventions: Biological: Red blood cell units stored >= 21 days

INTERVENTIONS:
Biological: Red blood cell units stored <= 10 days — Pre-storage leukoreduced red blood cell units stored <=10 days at time of transfusion. Can be AS1, AS3, or AS5. Frozen, deglycerolized, washed, and volume-reduced products are protocol violations.
  Arms: Shorter-storage red blood cell units
Biological: Red blood cell units stored >= 21 days — Pre-storage leukoreduced red blood cell units stored >=21 days at time of transfusion. Can be AS1, AS3, or AS5. Frozen, deglycerolized, washed, and volume-reduced products are protocol violations.
  Arms: Longer-storage red blood cell units

SUMMARY:
The RECESS study will compare the effects of transfusing red blood cell units stored <= 10 days vs. red blood cell units stored >= 21 days, in patients who are undergoing complex cardiac surgery and are likely to need a red blood cell transfusion. The primary hypothesis is that there is a clinically important difference between the effects of shorter-storage red cell units and longer-storage red cell units on clinical outcomes and mortality risk.

ELIGIBILITY:
Inclusion Criteria:

* >= 12 years old
* >= 40 kg body weight
* Scheduled complex cardiac surgery with planned use of median sternotomy.
* Patients ≥ 18 years must have a Transfusion Risk Understanding Scoring Tool (TRUST) probability score ≥ 3

Exclusion Criteria:

* Refusal of blood products
* Planned surgery is minimally invasive
* Known transfusion reaction history
* Requirement for washed products, volume reduced products, or products with additive solution removed
* Expected residual cyanosis with O2 saturation < 90
* Left ventricular assist device (LVAD) or Extracorporeal membrane oxygenation (ECMO) support pre-operatively or planned need post-operatively
* Cardiogenic shock requiring pre-operative placement of an Intra-aortic balloon pump (IABP) (IABP done for unstable angina or prophylactically for low ejection fraction is not excluded)
* Planned Deep Hypothermic Circulatory Arrest (DHCA)
* Renal dysfunction requiring pre-operative renal replacement therapies such as hemodialysis (HD) or continuous venovenous hemofiltration (CVVH)
* Planned use of alternative to heparin, e.g. bivalirudin
* Planned use of autologous or directed donations
* Prior RBC transfusion during hospitalization for the study-qualifying surgery
* Prior randomization into the RECESS study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1481 (Actual)
Dates: Start 2010-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F Assmann, PhD, Principal Investigator — Carelon Research; Steven Sloan, MD, Principal Investigator — Boston Children's Hospital; Thomas Ortel, MD, Principal Investigator — Duke University; Cassandra Josephson, MD, Principal Investigator — Emory University; Christopher Stowell, MD, Principal Investigator — Massachusetts General Hospital; Meghan Delaney, DO, Principal Investigator — University of Washington/Fred Hutchinson Cancer Research Center; Marie Steiner, MD, Principal Investigator — University of Minnesota Medical Center Fairview; Darrell Triulzi, MD, Principal Investigator — University of Pittsburgh Presbyterian and Shadyside; Lynne Uhl, MD, Principal Investigator — Beth Israel Deaconess Medical Center; Richard Kaufman, MD, Principal Investigator — Brigham and Women's Hospital; James Bussel, MD, Principal Investigator — Weill Medical College of Cornell University; Paul Ness, MD, Principal Investigator — Johns Hopkins University; Thomas Raife, MD, Principal Investigator — University of Iowa; Rhonda Cooke, MD, Principal Investigator — University of Maryland; Nigel Key, MD, Principal Investigator — University of North Carolina, Chapel Hill; Jeff Carson, MD, Principal Investigator — Rutgers, The State University of New Jersey; Vincent Scavo, MD, Principal Investigator — Indiana/Ohio Heart; Wade Fischer, MD, FACS, Principal Investigator — Froedtert Hospital; Pampee Young, MD, Principal Investigator — Vanderbilt University; Kathy Puca, MD, Principal Investigator — St. Luke's Hospital; James George, MD, Principal Investigator — University of Oklahoma; Gregory Nuttall, MD, Principal Investigator — Mayo Clinic; Arthur Bracey, MD, Principal Investigator — Texas Heart Institute; Richard Engleman, MD, Principal Investigator — Baystate Medical Center; Philip Greileich, MD, Principal Investigator — University of Texas; Kent Berg, MD, Principal Investigator — University of Florida; Robert Hunsaker, MD, Principal Investigator — St. Elizabeth's Medical Center; Ronald Miles, MD, Principal Investigator — Aspirus Medical Center; Ravindra Karanam, MD, Principal Investigator — Barnabas Health, Newark Beth Israel Medical Center; Cornelius Dyke, MD, Principal Investigator — Sanford Heart Center; Eldad Hod, MD, Principal Investigator — Columbia University Health Center
Locations (33):
- United States (33):
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - St. Joseph Hospital, Fort Wayne, Indiana
  - Indiana/Ohio Heart, Fort Wayne, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Fairview Southdale Hospital/University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Deaconess Medical Center, Newark, New Jersey
  - Columbia University Health Center, New York, New York
  - Weill Cornell Medical School, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Sanford Heart Center, Fargo, North Dakota
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Presbyterian and Shadyside, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - Veterans Administration Puget Sound, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
  - Aurora St. Lukes Medical Center, Milwaukee, Wisconsin
  - Aspirus Vascular Heart Center, Wausau, Wisconsin

REFERENCES:
- [Derived] Delaney M, Stark PC, Suh M, Triulzi DJ, Hess JR, Steiner ME, Stowell CP, Sloan SR. Massive Transfusion in Cardiac Surgery: The Impact of Blood Component Ratios on Clinical Outcomes and Survival. Anesth Analg. 2017 Jun;124(6):1777-1782. doi: 10.1213/ANE.0000000000001926. PMID 28333704
- [Derived] Steiner ME, Ness PM, Assmann SF, Triulzi DJ, Sloan SR, Delaney M, Granger S, Bennett-Guerrero E, Blajchman MA, Scavo V, Carson JL, Levy JH, Whitman G, D'Andrea P, Pulkrabek S, Ortel TL, Bornikova L, Raife T, Puca KE, Kaufman RM, Nuttall GA, Young PP, Youssef S, Engelman R, Greilich PE, Miles R, Josephson CD, Bracey A, Cooke R, McCullough J, Hunsaker R, Uhl L, McFarland JG, Park Y, Cushing MM, Klodell CT, Karanam R, Roberts PR, Dyke C, Hod EA, Stowell CP. Effects of red-cell storage duration on patients undergoing cardiac surgery. N Engl J Med. 2015 Apr 9;372(15):1419-29. doi: 10.1056/NEJMoa1414219. PMID 25853746
- [Derived] Kekre N, Mallick R, Allan D, Tinmouth A, Tay J. The impact of prolonged storage of red blood cells on cancer survival. PLoS One. 2013 Jul 16;8(7):e68820. doi: 10.1371/journal.pone.0068820. Print 2013. PMID 23874777
- [Derived] Berra L, Coppadoro A, Yu B, Lei C, Spagnolli E, Steinbicker AU, Bloch KD, Lin T, Sammy FY, Warren HS, Fernandez BO, Feelisch M, Dzik WH, Stowell CP, Zapol WM. Transfusion of stored autologous blood does not alter reactive hyperemia index in healthy volunteers. Anesthesiology. 2012 Jul;117(1):56-63. doi: 10.1097/ALN.0b013e31825575e6. PMID 22531338
- [Derived] Steiner ME, Assmann SF, Levy JH, Marshall J, Pulkrabek S, Sloan SR, Triulzi D, Stowell CP. Addressing the question of the effect of RBC storage on clinical outcomes: the Red Cell Storage Duration Study (RECESS) (Section 7). Transfus Apher Sci. 2010 Aug;43(1):107-16. doi: 10.1016/j.transci.2010.05.014. Epub 2010 Jul 23. PMID 20655807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: RECESS recruitment took place at 33 US hospitals, beginning in January 2010 and ending in January 2014.
Pre-assignment Details: Randomization was stratified by age (≥18 yrs or <18 yrs) and by whether or not the subject was in the ICU prior to surgery. A subject could not be randomized unless prior to surgery but no earlier than one calendar day prior to surgery, the transfusion service had enough suitable units of both storage durations to satisfy the cross-match request.
Period: Overall Study
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Started | 742 | 739
Completed | 538 | 560
Not Completed | 204 | 179
Not completed — no surgery w/in 30 days of randomization | 11 | 18
Not completed — Death | 3 | 0
Not completed — no RBCs received 96hrs after randomized | 186 | 155
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 3 | 4

BASELINE CHARACTERISTICS:
Population: Analysis is restricted to evaluable subjects (defined as randomized subjects who underwent cardiac surgery within 30 days after randomization and received at least one RBC transfusion between randomization and post-operative hour 96).
Groups:
- Total: Total of all reporting groups
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units | Total
Number analyzed (Participants) | 538 | 560 | 1098
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [66 to 80] | 72 [65 to 79] | 72 [66 to 79]
Age, Customized [Number; unit: participants]
  <18 years | 2 | 2 | 4
  >= 18 years | 536 | 558 | 1094
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 310 | 313 | 623
  Male | 228 | 247 | 475
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 19 | 32
  Not Hispanic or Latino | 506 | 513 | 1019
  Unknown or Not Reported | 19 | 28 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 11 | 8 | 19
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 32 | 39 | 71
  White | 485 | 493 | 978
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 4 | 15 | 19
Region of Enrollment [Number; unit: participants]
  United States | 538 | 560 | 1098
Weight [Median (Inter-Quartile Range); unit: kg] | 75 [65 to 89] | 74 [66 to 86] | 75 [66 to 87]
Height [Median (Inter-Quartile Range); unit: cm] | 165 [158 to 173] | 165 [160 to 175] | 165 [158 to 173]
Minimum TRUST Score [Number; unit: participants] — Per Alghamdi et al article in Transfusion (2006), the Transfusion Risk Understanding Scoring Tool (TRUST) score is an additive algorithm that provides an overall score that ranges from 0 to 8. The interpretation of the total score as it relates to the probability of exposure to transfusion is as follows: 0=baseline risk; 1=low risk; 2=intermediate risk; 3=high risk; 4-8=very high risk.
  participants
    0 | 1 | 0 | 1
    3 | 166 | 222 | 388
    4 | 210 | 196 | 406
    5 | 132 | 113 | 245
    6 | 26 | 27 | 53
    7 | 3 | 2 | 5
ICU Status at Randomization [Number; unit: participants]
  In ICU Before Surgery | 34 | 33 | 67
  Not in ICU Before Surgery | 504 | 527 | 1031
Baseline Multiple Organ Dysfunction Score [Number; unit: participants] — Per Marshall et al article in Critical Care Medicine (1995), increasing Multiple Organ Dysfunction Scores correlated with in-hospital mortality. No deaths occurred in patients with a MODS score of 0. The approximate in-hospital mortality rates were 6% for patients with MODS score of 1-4 points, 15% for patients with scores between 5-8, 50% for patients with scores between 8-12, 68% for patients with scores 13-16, 80% for patients with scores 17-20 and 100% for scores > 20.
  participants
    0 | 252 | 293 | 545
    1 | 223 | 194 | 417
    2 | 48 | 57 | 105
    3 | 10 | 11 | 21
    4 | 4 | 4 | 8
    5 | 1 | 1 | 2
ABO Blood Group [Number; unit: participants]
  O | 209 | 235 | 444
  A | 240 | 241 | 481
  B | 64 | 63 | 127
  AB | 25 | 21 | 46
Hemoglobin [Median (Inter-Quartile Range); unit: g/L] | 11.7 [10.7 to 12.8] | 12.0 [10.8 to 13.0] | 11.9 [10.7 to 12.9]

OUTCOME MEASURES:

1. Primary Outcome: The Change in the Composite Multiple Organ Dysfunction Score (MODS) From the Pre-operative Baseline. The Worst Post-operative Values of Each Component of MODS Will be Used to Calculate the Change in MODS.
Description: The follow-up MODS used to calculate 7-day ΔMODS from pre-op baseline was based on the worst value of each component of MODS observed through post-op day 7, hospital discharge, or death, whichever occurred first, even if a subject's worst values for different components occurred on different dates. Subjects who died during this time period were assigned the worst possible follow-up MODS score, 24 points, and each component of MODS was set at 4, which is the worst score. If a subject did not die during this time period but had at least one day where the Glasgow Coma Score couldn't be scored [subject sedated; neurologic function not normal by pre-op history (prior stroke, tumor or trauma sequelae, cognitively challenged, behavioral disorder, etc.) or intra-op history, but currently unable to assess because of sedation], then a post-op MODS score was set to missing and a 7-day ΔMODS was not computed. The total MODS score ranges from 0 (best possible) to 24 points (worst possible).
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: MOD score points
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 534 | 553
MOD score points | 8.49 (3.62) | 8.66 (3.55)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.44, ANCOVA; The treatment groups were compared with respect to the change in MODS, adjusting for baseline MODS; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.60 to 0.26] — The longer storage red blood cell units arm is the reference category. After adjusting for baseline MODS, the difference in the means was -0.17, positive values are in favor of longer storage duration

2. Secondary Outcome: All-cause Mortality
Description: Subjects were randomized for RECESS no earlier than one calendar day before the planned date of surgery, and were followed for all-cause mortality until post-operative Day 28, death, or study withdrawal, whichever occurred first. In some cases the surgery was postponed after randomization had already occurred. If surgery did not occur within 30 days after randomization, the subject ended the study and was not considered evaluable. If surgery did occur within 30 days after randomization, and the subject received at least one RBC transfusion between randomization and 96 hours after the end of surgery, the subject was considered evaluable. Therefore, in a few evaluable subjects, post-operative Day 28 could be nearly two months after the date of randomization. The times in the time-to-event analysis started at randomization.
Time Frame: 28 days post-surgery
Population: as for baseline characteristics
Measure: Number; unit: participants with event
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 538 | 560
participants with event | 23 | 29
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.50, Regression, Cox; The treatment groups were compared with respect to all-cause mortality, adjusting for baseline MODS; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.48 to 1.43] — The longer storage duration arm is the reference category

3. Secondary Outcome: Change in Multiple Organ Dysfunction Score From Pre-operative Baseline.
Description: The follow-up MODS used to calculate 28-day ΔMODS from pre-op baseline was based on the worst value of each component of MODS observed through post-op day 28, hospital discharge, or death, whichever occurred first, even if a subject's worst values for different components occurred on different dates. Subjects who died during this time period were assigned the worst possible follow-up MODS score, 24 points, and each component of MODS was set at 4, which is the worst score. If a subject did not die during this time period but had at least one day where the Glasgow Coma Score couldn't be scored[subject sedated; neurologic function not normal by pre-op history (prior stroke, tumor or trauma sequelae, cognitively challenged, behavioral disorder, etc.) or intra-op history, but currently unable to assess because of sedation], then a post-op MODS score was set to missing and a 28-day ΔMODS was not computed. The total MODS score ranges from 0 (best possible) to 24 points (worst possible).
Time Frame: Through 28 days post-surgery, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: MOD score points
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 531 | 555
MOD score points | 8.74 (4.04) | 9.07 (4.22)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.20, ANCOVA; The treatment groups were compared with respect to 28-day change in MODS, adjusting for baseline MODS; Mean Difference (Net) = -0.32, 95% CI 2-sided [-0.82 to 0.17] — The longer storage red blood cell units arm is the reference category. After adjusting for baseline MODS, the difference in the means was -0.32; positive values are in favor of longer storage duration

4. Secondary Outcome: Composite of Major In-hospital Post-operative Complications (Death, Stroke, Myocardial Infarction, Renal Failure, Culture-proven Sepsis/Septic Shock)
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Number; unit: participants with event
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 448 | 470
participants with event | 91 | 87
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.50, Fisher Exact; Risk Difference (RD) = 0.018, 95% CI 2-sided [-0.033 to 0.069] — The difference in proportions between the two treatment arms was computed as the proportion of subjects with the event in the shorter storage duration arm minus the proportion of subjects with the event in the longer storage duration arm

5. Secondary Outcome: Composite of Major Cardiac Events (Death, Myocardial Infarction, Low Cardiac Output, Ventricular Tachycardia, Ventricular Fibrillation)
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Number; unit: participants with event
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 472 | 496
participants with event | 206 | 230
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.40, Fisher Exact; Risk Difference (RD) = -0.027, 95% CI 2-sided [-0.090 to 0.035] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Composite of Major Pulmonary Events (Any Mechanical Ventilation From 48 Hours Post-operation to Day 7, Hospital Discharge or Death, Whichever Comes First, or Pulmonary Embolism)
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Number; unit: participants with event
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 508 | 537
participants with event | 62 | 75
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.41, Fisher Exact; Risk Difference (RD) = -0.018, 95% CI 2-sided [-0.059 to 0.023] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Ventilation Duration
Description: Because some subjects may experience multiple periods of ventilator use, the total duration that they were on a ventilator was compared between the two groups.
Time Frame: Through post-operative day 28, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 514 | 540
days | 2.7 (3.9) | 2.8 (4.3)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.75, Kruskal-Wallis; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.62 to 0.37]

8. Secondary Outcome: Change in Serum Creatinine From Pre-operative Value to Worst Post-operative Value
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 532 | 558
mg/dL | 0.35 (0.58) | 0.35 (0.51)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.62, ANCOVA; The treatment arms were compared with respect to the change in creatinine, adjusting for the baseline creatinine value; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.08 to 0.05] — The longer storage red blood cell units arm is the reference category. After adjusting for baseline creatinine, the difference in the means was -0.02, positive values are in favor of longer storage duration

9. Secondary Outcome: Change in Troponin-I From Pre-operative Value to Worst Post-operative Value
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 443 | 470
ng/mL | 15.82 (37.64) | 14.06 (23.77)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Troponin-I values recorded as 'too low to detect' were recoded as 0 since the median value of the minimum quantitative troponin-I value obtained among all participating sites was 0.01; Test type: Superiority or Other; p = 0.35, ANCOVA — The treatment arms were compared with respect to the change in troponin-I, adjusting for the baseline troponin-I value; Mean Difference (Net) = 1.93, 95% CI 2-sided [-2.11 to 5.98] — The longer storage red blood cell units arm is the reference category. After adjusting for baseline troponin-I, the change in troponin-I values was 1.9 ng/mL higher in the shorter storage red blood cell units arm

10. Secondary Outcome: Change in Lactate From Pre-operative Value to Worst Post-operative Value
Description: The arterial lactate levels were adjusted to make them comparable to venous lactate levels.
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 410 | 437
mmol/L | 2.30 (3.33) | 2.92 (5.97)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.10, Kruskal-Wallis

11. Secondary Outcome: Change in Bilirubin From Pre-operative Value to Worst Post-operative Value
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 513 | 543
mg/dL | 0.85 (1.24) | 1.49 (2.53)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p < 0.01, ANCOVA; Mean Difference (Net) = -0.65, 95% CI 2-sided [-0.89 to -0.41] — The longer storage red blood cell units arm is the reference category. After adjusting for baseline bilirubin, the change in bilirubin values was 0.65 mg/dL lower in the shorter storage red blood cell units arm

12. Secondary Outcome: Change in ALT From Pre-operative Value to Worst Post-operative Value (for Pediatric Subjects Only)
Time Frame: Through post-operative day 7, hospital discharge, or death, whichever occurs first
Population: Only 4 pediatric subjects were enrolled. One treatment arm had only one subject with available data for analyzing the change in ALT. Therefore, to protect patient confidentiality, results were not entered.
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Days to First Bowel Movement
Description: Subjects were randomized for RECESS no earlier than one calendar day before the planned date of surgery, and were followed until post-operative Day 28, death, or study withdrawal, whichever occurred first. In some cases the surgery was postponed after randomization had already occurred. If surgery did not occur within 30 days after randomization, the subject ended the study and was not considered evaluable. If surgery did occur within 30 days after randomization, and the subject received at least one RBC transfusion between randomization and 96 hours after the end of surgery, the subject was considered evaluable. Therefore, in a few evaluable subjects, post-operative Day 28 could be nearly two months after the date of randomization. The times in the time-to-event analyses are from randomization to first post-operative bowel movement.
Time Frame: Through post-operative day 28, hospital discharge, or death, whichever occurs first
Population: Analysis is restricted to evaluable subjects (defined as randomized subjects who underwent cardiac surgery within 30 days after randomization and received at least one RBC transfusion between randomization and post-operative hour 96). The mean time to an event is estimated by the area under the survival function.
Measure: Mean (Standard Error); unit: days
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 538 | 560
days | 5.89 (0.17) | 6.62 (0.25)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.11, Regression, Cox — The treatment groups were compared with respect to days to first post-operative bowel movement, adjusting for baseline MODS; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.98 to 1.25] — The longer storage duration arm is reference category

14. Secondary Outcome: Days to First Solid Food
Description: Subjects were randomized for RECESS no earlier than one calendar day before the planned date of surgery, and were followed until post-operative Day 28, death, or study withdrawal, whichever occurred first. In some cases the surgery was postponed after randomization had already occurred. If surgery did not occur within 30 days after randomization, the subject ended the study and was not considered evaluable. If surgery did occur within 30 days after randomization, and the subject received at least one RBC transfusion between randomization and 96 hours after the end of surgery, the subject was considered evaluable. Therefore, in a few evaluable subjects, post-operative Day 28 could be nearly two months after the date of randomization. The times in the time-to-event analyses are from randomization to first post-operative solid food.
Time Frame: Through post-operative day 28, hospital discharge, or death, whichever occurs first
Population: as for outcome 13
Measure: Mean (Standard Error); unit: days
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 538 | 560
days | 5.73 (0.37) | 6.18 (0.35)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.22, Regression, Cox; The treatment groups were compared with respect to days to first post-operative solid food, adjusting for baseline MODS; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.96 to 1.22] — The longer storage duration arm is reference category

15. Secondary Outcome: Days Alive and Ventilator Free Through Post-op Day 28
Time Frame: Through post-op day 28
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 511 | 539
days | 25.38 (6.40) | 25.17 (6.75)
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.71, Kruskal-Wallis; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.59 to 1.00] — The longer storage duration arm is reference category

16. Secondary Outcome: Any Mechanical Ventilation More Than 48 Hours Post-operation
Time Frame: 48 hours post-operation through day 28, hospital discharge, or death, whichever occurs first
Population: as for baseline characteristics
Measure: Number; unit: participants with event
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Number analyzed (Participants) | 508 | 537
participants with event | 68 | 80
Statistical Analysis 1: Comparison: Shorter-storage Red Blood Cell Units vs Longer-storage Red Blood Cell Units; Test type: Superiority or Other; p = 0.53, Fisher Exact; Risk Difference (RD) = -0.015, 95% CI 2-sided [-0.057 to 0.027] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include any untoward medical occurrence which occurred after a subject gave informed consent and no later than post-operative day 28, hospital discharge, or death, whichever came first.
Description: Data were collected on all serious adverse events (SAEs) and on pre-specified types of non-serious adverse events. If a subject experiences more than one occurrence of a specific adverse event, the subject was counted only once for that adverse event.
Arm/Group | Shorter-storage Red Blood Cell Units | Longer-storage Red Blood Cell Units
Serious Adverse Events (participants affected / at risk) | 283/538 | 288/560
Other Adverse Events (participants affected / at risk) | 324/538 | 334/560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shorter-storage Red Blood Cell Units (N=538) | Longer-storage Red Blood Cell Units (N=560)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 7 (7) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Accelerated idioventricular rhythm (Cardiac disorders) | 3 (4) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 9 (9) | 9 (9)
Acute right ventricular failure (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 31 (33) | 25 (28)
Atrial flutter (Cardiac disorders) | 3 (3) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 7 (9) | 10 (10)
Cardiac arrest (Cardiac disorders) | 3 (4) | 4 (4)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac tamponade (Cardiac disorders) | 6 (6) | 5 (6)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 9 (9) | 13 (13)
Cardiomyopathy acute (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Negative cardiac inotropic effect (Cardiac disorders) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 20 (20) | 24 (24)
Sinus tachycardia (Cardiac disorders) | 16 (17) | 26 (28)
Supraventricular tachyarrhythmia (Cardiac disorders) | 3 (3) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Tachycardia (Cardiac disorders) | 0 (0) | 5 (6)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular asystole (Cardiac disorders) | 2 (2) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 4 (4) | 6 (6)
Ventricular tachyarrhythmia (Cardiac disorders) | 3 (4) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 6 (9) | 7 (8)
Familial hypocalciuric hypercalcaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Heart block congenital (Congenital, familial and genetic disorders) | 1 (1) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Antidiuretic hormone abnormality (Endocrine disorders) | 1 (1) | 0 (0)
Visual acuity reduced transiently (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Megacolon (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesenteric occlusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Application site bleeding (General disorders) | 13 (13) | 11 (11)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Infusion site dermatitis (General disorders) | 0 (0) | 1 (1)
Multi-organ disorder (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 26 (28) | 51 (58)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactoid shock (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (2) | 2 (2)
Abdominal sepsis (Infections and infestations) | 0 (0) | 2 (2)
Acute endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Adenoviral upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 3 (3) | 6 (6)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 11 (12) | 9 (9)
Candida pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 3 (3) | 3 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 3 (3)
Genitourinary tract infection (Infections and infestations) | 8 (9) | 6 (6)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 2 (2)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Serratia infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Confusion postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative renal failure (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Procedural hypotension (Injury, poisoning and procedural complications) | 3 (3) | 9 (9)
Renal injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 10 (10) | 10 (10)
Weaning failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time (Investigations) | 0 (0) | 1 (1)
Anticoagulation drug level below therapeutic (Investigations) | 1 (1) | 0 (0)
Aspiration pleural cavity (Investigations) | 1 (1) | 1 (1)
Bacteria blood identified (Investigations) | 1 (1) | 0 (0)
Bacteria sputum identified (Investigations) | 0 (0) | 1 (1)
Blood gases abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 6 (6) | 5 (5)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0)
Blood urea nitrogen/creatinine ratio increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 1 (1)
Body temperature decreased (Investigations) | 2 (2) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 3 (3)
Bronchoalveolar lavage abnormal (Investigations) | 0 (0) | 1 (1)
Cardiac enzymes increased (Investigations) | 2 (2) | 2 (2)
Cardiac output decreased (Investigations) | 1 (1) | 0 (0)
Clostridium difficile toxin test positive (Investigations) | 0 (0) | 1 (1)
ECG signs of myocardial ischaemia (Investigations) | 4 (4) | 2 (2)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Fungus culture positive (Investigations) | 1 (1) | 0 (0)
Heart rate decreased (Investigations) | 0 (0) | 2 (2)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio abnormal (Investigations) | 1 (1) | 0 (0)
Kidney injury molecule-1 (Investigations) | 1 (1) | 1 (1)
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 0 (0) | 1 (1)
NIH stroke scale (Investigations) | 1 (1) | 0 (0)
NIH stroke scale score increased (Investigations) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 1 (2)
Oxygen saturation (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 2 (2) | 1 (1)
Pathology test (Investigations) | 0 (0) | 1 (1)
Radial pulse abnormal (Investigations) | 0 (0) | 1 (1)
Red blood cells urine positive (Investigations) | 1 (1) | 0 (0)
Sputum culture positive (Investigations) | 1 (1) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 1 (1)
Troponin I increased (Investigations) | 2 (2) | 0 (0)
Urine output decreased (Investigations) | 15 (15) | 18 (18)
White blood cell count increased (Investigations) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 7 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 15 (15) | 15 (16)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 55 (56) | 46 (52)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Anoxic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Atonic seizures (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 5 (5) | 3 (3)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 5 (5) | 2 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Seizure anoxic (Nervous system disorders) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 15 (16) | 14 (14)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemoglobinuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Oliguria (Renal and urinary disorders) | 5 (5) | 3 (3)
Renal disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 5 (5)
Renal failure acute (Renal and urinary disorders) | 8 (8) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2) | 3 (3)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 5 (5)
Bleeding anovulatory (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 11 (11)
Anaemic hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6)
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Clotted haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 24 (25)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 12 (12)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 33 (36) | 39 (39)
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 9 (9)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax spontaneous tension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 12 (12)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Abdominal exploration (Surgical and medical procedures) | 1 (1) | 0 (0)
Allergy prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)
Aneurysm repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Dialysis (Surgical and medical procedures) | 0 (0) | 1 (1)
Extracorporeal membrane oxygenation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotensive anaesthesia procedure (Surgical and medical procedures) | 3 (3) | 2 (2)
Incisional drainage (Surgical and medical procedures) | 2 (2) | 2 (2)
Intracerebral haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1)
Pericardial drainage (Surgical and medical procedures) | 1 (1) | 0 (0)
Removal of foreign body (Surgical and medical procedures) | 1 (1) | 0 (0)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (2)
Accelerated hypertension (Vascular disorders) | 2 (2) | 1 (1)
Aortic intramural haematoma (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Diastolic hypertension (Vascular disorders) | 0 (0) | 2 (2)
Diastolic hypotension (Vascular disorders) | 14 (14) | 14 (14)
Essential hypertension (Vascular disorders) | 5 (5) | 3 (3)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 13 (14) | 13 (13)
Hypotension (Vascular disorders) | 97 (106) | 87 (96)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 2 (2)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (1)
Labile hypertension (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shorter-storage Red Blood Cell Units (N=538) | Longer-storage Red Blood Cell Units (N=560)
Haemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 7 (7) | 4 (4)
Accessory cardiac pathway (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 10 (10)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 12 (12) | 11 (12)
Sinus tachycardia (Cardiac disorders) | 25 (27) | 28 (28)
Supraventricular tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachyarrhythmia (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 7 (7) | 3 (3)
Familial hypocalciuric hypercalcaemia (Congenital, familial and genetic disorders) | 4 (4) | 2 (2)
Adverse reaction (General disorders) | 0 (0) | 1 (1)
Catheter site phlebitis (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 78 (89) | 98 (107)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Alloimmunisation (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Acinetobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Actinomycotic pulmonary infection (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Application site cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 1 (1)
Aspergillosis oral (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 2 (2)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Genitourinary tract infection (Infections and infestations) | 10 (10) | 9 (10)
Incision site infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 2 (2)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Iatrogenic injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Urethral stricture traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 7 (7) | 10 (10)
Bacteria blood identified (Investigations) | 0 (0) | 1 (1)
Bacteria sputum identified (Investigations) | 2 (2) | 1 (1)
Bacteria urine (Investigations) | 1 (1) | 0 (0)
Bilirubin conjugated abnormal (Investigations) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 2 (2)
Blood pressure abnormal (Investigations) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 5 (5) | 3 (3)
Blood pressure orthostatic decreased (Investigations) | 1 (1) | 0 (0)
Blood urine (Investigations) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 8 (8) | 3 (3)
Cardiac enzymes increased (Investigations) | 7 (7) | 9 (9)
Differential white blood cell count normal (Investigations) | 0 (0) | 1 (1)
ECG signs of myocardial ischaemia (Investigations) | 7 (7) | 8 (8)
Heart rate decreased (Investigations) | 1 (1) | 0 (0)
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Sputum culture (Investigations) | 1 (1) | 0 (0)
Sputum culture positive (Investigations) | 2 (3) | 0 (0)
Troponin (Investigations) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 3 (3) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 18 (18) | 18 (18)
Hyperphosphataemia (Metabolism and nutrition disorders) | 25 (30) | 11 (13)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 187 (230) | 191 (228)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 8 (8) | 5 (7)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Haemoglobinuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hypocalciuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Oliguria (Renal and urinary disorders) | 2 (2) | 4 (4)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal impairment (Renal and urinary disorders) | 2 (2) | 2 (3)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary retention (Renal and urinary disorders) | 5 (5) | 3 (3)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anaemic hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 11 (11)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 20 (20)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 14 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 12 (12)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Haemophilus influenzae type b immunisation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotensive anaesthesia procedure (Surgical and medical procedures) | 1 (1) | 1 (1)
Accelerated hypertension (Vascular disorders) | 4 (4) | 5 (5)
Diastolic hypertension (Vascular disorders) | 2 (3) | 1 (1)
Diastolic hypotension (Vascular disorders) | 6 (6) | 4 (4)
Essential hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 20 (20) | 21 (23)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 71 (76) | 73 (76)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Only 4 pediatric subjects were enrolled. One treatment arm had only one subject with available data for analyzing the change in ALT outcome. Therefore, to protect patient confidentiality, results were not entered for this outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No